CLINICAL TRIAL: NCT03936387
Title: Bilateral Continuous Erector Spinae Blocks for Post-Sternotomy Pain Management: A Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Roland Brusseau, SeniorAssociate in Perioperative Anesthesia, Department of Anesthesiology, Perioperative and Pain Medicine Instructor in Anaesthesia, Harvard Medical School, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00031524
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Pain, Postoperative
Keywords: erector spinae block; regional anesthesia; sternotomy; ropivacaine
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Single intervention group, bilateral erector spinae blocks with 0.2% ropivacaine, to assess the feasibility of this technique for postoperative pain control following surgeries involving sternotomies in children.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Bilateral erector spinae blocks (Experimental): Bilateral erector spinae block catheters are placed at end of the sternotomy procedure, bolused with 1ml/kg 0.2% ropivacaine, then started on a 0.2ml/kg/hour continuous infusion of 0.2% ropivacaine. Patients will have access to rescue opiates as needed by means of the standard PCA/NCA demand protocols utilized at BCH.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Erector spinae blocks: T4/5 transverse process is identified with the ultrasound transducer in a parasagittal orientation; the needle tip is advanced until it contacts the transverse process, just below the erector spinae muscle complex; the erector spinae muscle is visualized to be elevated up off of the transverse process with normal saline injection. Following a bolus injection of 2ml/kg of 0.2% ropivacaine, a catheter is threaded into the space occupied by the local anesthetic bolus. Repeated on contralateral side.
  Other Names: Naropin

SUMMARY:
Overall Aim: To evaluate the feasibility and potential benefits of investigating bilateral continuous erector spinae blocks (BESB) for postoperative pain management in a small cohort of children undergoing surgical sternotomy prior to planning an appropriately powered, randomized, controlled trial of the same.

Hypothesis: The investigators' primary hypothesis is that utilizing bilateral erector spinae blocks for post-sternotomy pain is a feasible intervention for consideration in a larger trial by demonstrating a 75% or greater successful intervention completion rate without any major adverse outcomes.

DETAILED DESCRIPTION:
Regional anesthesia-and pediatric regional anesthesia in particular-is a rapidly evolving subfield of anesthesia practice driven with considerable urgency by the growing recognition that even appropriate perioperative narcotic administration can have significant derogatory long-term effects.

Regional anesthetics can provide targeted, continuous analgesia to select dermatomes with minimal additional patient risk and as such have become routine components of opioid-sparing intraoperative and postoperative pain management plans for surgical patients at BCH. In addition to the postulated benefit of reducing overall opioid exposure and potentially reducing the risk for long term physiologic and behavioral dependence upon opioids, regional anesthetics may allow for earlier extubation after selected surgeries, shorter ICU, PACU and inpatient admissions, earlier mobilization, fewer gastrointestinal complications, and improved patient satisfaction scores.

Despite a robust literature supporting the safety and efficacy of regional anesthesia for postoperative pain control across a broad range or surgery types, patient demographics and underlying comorbidities, there are certain classes of surgeries that have (to date) not benefitted from the advantages that regional anesthetics may provide, most notably spine surgery and cardiac surgery.

Concerns have been expressed with regard to regional anesthetics for cardiac surgeries in particular (this being the primary surgical type associated with sternotomies in a pediatric populations), given that most patients are pharmacologically anticoagulated to some extent during their procedures and are thus at increased risk for bleeding. This is further complicated in the pediatric cardiac surgical population as many of these children are intubated for an extended period of time and therefore may not have particularly reliable neurological exams in the setting of neuraxial regional anesthetics-potentially resulting in unrecognized acquired neurological defecits. While there is emerging evidence of improved outcomes with neuraxial regional anesthetics in adult cardiac surgery patients, this has not trickled down to the pediatric population, likely for some of these reasons.

The investigators at BCH are fortunate to have one of the largest concentrated pediatric cardiac surgical populations in the US along with an active, and well organized regional anesthesia service. Because of this, the investigators are in a unique position to more thoroughly evaluate the effectiveness and safety of regional anesthetics in children following cardiac surgery. Furthermore it is thought to be critical that institutions such as BCH take a leading role in documenting the effects of regional anesthesia on the most important outcome measures when considering perioperative medicine. These include: overall pain management, surgical healing, functional recovery, long term pain symptoms, and emotional/behavioral outcomes after surgery.

Recently, the erector spinae block (ESB) has become popular for providing analgesia after a number of anterior chest and abdominal procedures. This is a simple interfascial plane block that can reliably provide unilateral chest and/or abdominal wall analgesia. It has been described in numerous case reports and one case series as an effective block for management of unilateral thoracotomies, unilateral rib fractures, unilateral abdominal incisions and most notably, when used bilaterally, for management of post-sternotomy pain. New case reports and series involving the ESB are being published almost weekly at this point with a growing literature specific to cardiac surgical applications. Indeed a randomized controlled trial to investigate the analgesic efficacy of bilateral erector spinae plane (BESP) blocks compared with conventional treatment for pain after cardiac surgery in adult patients was published recently (2018) with promising results.

As an interfascial plane block in a compressible anatomical space, the ESB is thought to be safe in anticoagulated (or recently anticoagulated) patients. It is fast becoming a preferred anesthetic option for these pharmacologically or otherwise coagulopathic patients as opposed to neuraxial (e.g. epidural) and paraneuraxial blocks (i.e. paravertebral) nerve blocks, which are largely contraindicated in this setting.

Given the ESB's potentially favorable risk profile versus the other blocks that would subserve the same dermatomes (i.e. it is technically less challenging, more distant from critical structures, and thought to be safe in anticoagulated patients) it could provide both a safer and easier to perform regional anesthesia option for many patients. In particular, it offers a new option for a subset of anticoagulated patients for whom other regional techniques (epidural, paravertebral) are contraindicated. This is particularly true for the populations of pediatric cardiac surgical patients at BCH if used bilaterally.

Indeed, given the current information available related to the ESB, the regional anesthesia service at BCH has begun employing it when possible in circumstances when a neuraxial or paravertebral block(s) would commonly be used but is/are relatively or absolutely contraindicated. Patients undergoing thoracotomies while anticoagulated for cardiopulmonary bypass, aortic clamping, etc. have been successfully managed with unilateral continuous ESBs. In addition, thoracotomies in patients with acquired (e.g. dilutional) and other pathologic coagulopathies have been managed with ESBs. As such, the ESB has been adopted for routine use in specific patient populations at BCH and has even occasionally been utilized in lieu of the more longstanding routine PVBs or epidural blocks for patients without contraindication for such.

Retrospective review of BCH outcomes data for 67 ESBs done for a variety of surgeries and populations has not revealed any significant differences between PVBs and ESBs in terms of adverse events, postoperative opiate use, median pain scores, or other standard outcomes measures. As this data is observational in nature, it is difficult to draw firm conclusions as to the efficacy of the two blocks. However, since there are distinct known and described advantages associated with regional anesthetics for postoperative pain management, it would be prudent to evaluate these blocks in a controlled, randomized, trial. Prior to such a trial, a pilot study to evaluate the feasibility of such a trial is warranted.

As such, the investigators propose to evaluate the feasibility of investigating bilateral continuous erector spinae blocks (BESB) for patients undergoing surgical sternotomy by means of a pilot study. For this study, 'feasibility' will be defined primarily as a successful intervention completion rate of 75% or greater of all subjects with no major adverse outcomes. Secondary measures of feasibility will include aggregate 'data integrity' as defined by successful collection of 75% or greater of all possible data points for successfully completed subjects as well as 'efficient intervention duration' as evaluated by intervention completion time being less than 40 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled as part of the cardiac surgical ERAS program.
2. Scheduled for a primary sternotomy.
3. Ages 3-21 years.

Exclusion Criteria:

1. Patients undergoing reoperative procedures.
2. Significant scoliosis or other anatomic contraindications to ESB.
3. History of bleeding or current therapeutic dose anticoagulant use.
4. Significant intraoperative hemodynamic instability or bleeding, as ascertained by clinicians taking care of the patient.
5. Patients with severe neurodevelopmental delays.
6. Patients with previous chronic pain syndromes.
7. Patients with a history of opioid treatment at any point in the 2 months prior to surgery.
8. Lack of parental consent and/or child assent.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ROLAND BRUSSEAU, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children"S Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bilateral Erector Spinae Blocks
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 9.0 [5.2 to 12.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Completed a Successful Intervention With No Major Adverse Events
Description: For this study, 'feasibility' will be defined primarily as a successful intervention completion rate of 75% or greater of all subjects with no major adverse outcomes.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 10
Participants | 10

2. Secondary Outcome: Number of Participants Who Completed a Successful Intervention With a Full Data Set
Description: Secondary measures of feasibility will include aggregate 'data integrity' as defined by successful collection of 75% or greater of all possible data points for successfully completed subjects as well as 'efficient intervention duration' as evaluated by intervention completion time being less than 40 minutes.
Time Frame: 48 hours
Measure: Number; unit: participants
Arm/Group | Bilateral Erector Spinae Blocks
Number analyzed (Participants) | 10
participants | 10

ADVERSE EVENTS:
Time Frame: Until the first postoperative visit (usually one-month postop).
Arm/Group | Bilateral Erector Spinae Blocks
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT03936387/Prot_SAP_001.pdf